CLINICAL TRIAL: NCT02467322
Title: To Study The Incidence And Outcome Of Paracentesis Induced Circulatory Dysfunction In Decompensated Cirrhotics Undergoing Less Than 5 Litres Of Ascitic Fluid Tap With Or Without Albumin Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-003
Record Dates: First submitted 2015-06-04; First posted 2015-06-10 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2016-10

CONDITIONS: Decompensated Cirrhosis
MeSH Terms: interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albumin (Experimental): MVP (Moderate Volume Paracentesis) of less than 5 liters with iv albumin at a dose 8 gms/l of ascitic fluid.
  Interventions: Drug: Albumin; Drug: ascitic fluid
- No Albumin (Active Comparator): MVP(Moderate Volume Paracentesis) of less than 5 liters without albumin.
  Interventions: Drug: ascitic fluid

INTERVENTIONS:
Drug: Albumin — MVP of less than 5 liters with iv albumin at a dose 8 gms/L of ascitic fluid.
  Arms: Albumin
Drug: ascitic fluid

SUMMARY:
All consecutive patients admitted in ILBS from MAY 2015 to DECEMBER 2016. Decompensated cirrhosis patients will be randomized into Group 1: MVP (Moderate Volume Paracentesis) of less than 5 litres with iv albumin at a dose 8 gms/l of ascitic fluid Group 1: MVP (Moderate Volume Paracentesis) of less than 5 litres without albumin .

ELIGIBILITY:
Inclusion Criteria:

1. All Cirrhotics decompensated with ascites admitted in the hospital.
2. Grade II/III ascites
3. Need for paracentesis.

Exclusion Criteria:

1. Age <12 or > 75 years
2. Hepatocellular carcinoma
3. Non cirrhotic ascites such as malignancy or tubercular peritonitis
4. Serum Cr >1.5mg%
5. Refractory septic shock
6. Grade III/IV hepatic encephalopathy
7. Abdominal wall cellulitis
8. Active variceal bleed
9. Respiratory, cardiac and renal failure
10. Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of PICD (Paracentesis Induced Circulatory Dysfunction). | 1 Year

SECONDARY OUTCOMES:
Survival | 28 days
Total number of patients develop Hepatorenal Syndrome. | 1 Year
Total number of patients develop hyponatremia. | 1 Year
Changes in plasma Renin activity. | 1 Year
Changes in aldosterone with volume of ascitic fluid tap. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India